CLINICAL TRIAL: NCT04201964
Title: Improving Neuroprotective Strategy for Ischemic Stroke With Poor Recanalization After Thrombectomy by Intra-arterial TNK (INSIST-TNK): a Prospective, Single Arm, Pilot Study
Brief Title: Improving Neuroprotective Strategy for Ischemic Stroke With Poor Recanalization After Thrombectomy by Intra-arterial TNK (INSIST-TNK)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k(2019)30
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-arterial administration of tenecteplase (Experimental): Intra-arterial administration of tenecteplase (0.2-0.4 mg/min) immediately after thrombectomy device pass for 30-40 minutes.
  Interventions: Drug: Intra-arterial administration of tenecteplase

INTERVENTIONS:
Drug: Intra-arterial administration of tenecteplase — Intra-arterial administration of tenecteplase (0.2-0.4 mg/min) immediately after thrombectomy device pass for 30-40 minutes.

SUMMARY:
In 2015, five randomized trials showed efficacy of endovascular thrombectomy over standard medical care in patients with acute ischemic stroke caused by occlusion of arteries of the proximal anterior circulation. However, sufficient recanalization (mTICI2b-3) can 't be acquired in all patients under thrombectomy. There is a lack of evidence that whether salvage intra-arterial thrombolysis is beneficial for patients with insufficient recanalization after endovascular thrombectomy. The EXTEND-IA TNK study indicated that tenecteplase before thrombectomy was associated with a higher incidence of reperfusion and better functional outcome than alteplase among patients with ischemic stroke treated within 4.5 hours after symptom onset. This study intends to explore the proportion of sufficient recanalization (2b/3) after intra-arterial tenecteplase administration in patients undergoing thrombectomy with insufficient recanalization (1/2a).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients who presented with acute ischemic stroke and a large vessel occlusion in the anterior circulation and met the criteria of mechanical thrombectomy;
3. insufficient perfusion (mTICI 1/2a) after endovascular treatment;
4. The availability of informed consent.

Exclusion Criteria:

1. Sufficient recanalization (TICI 2b-3);
2. More than 3 times of thrombectomy device passes
3. Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage
4. Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia ( <100000/mm3)
5. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis
6. Severe uncontrolled hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg)
7. Patients allergic to any ingredient of drugs in our study
8. Unsuitable for this clinical studies assessed by researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of sufficient recanalization | immediately after local TNK treatment
  sufficient recanalization is defined as TICI 2b-3

SECONDARY OUTCOMES:
Proportion of favorable outcome | 90 days
  favorable outcome is defined as mRS 0-2
proportion of early neurological improvement | 48 hours
  early neurological improvement is defined as more than 4 decrease in NIHSS

OTHER OUTCOMES:
incidence of symptomatic intracranial haemorrhage | 48 hours
  intracranial haemorrhage is defined as more than 4 increase in NIHSS caused by intracranial bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China